CLINICAL TRIAL: NCT03722914
Title: A Multicentric Randomized Double-blind Placebo-controlled Study on the Efficacy and Safety of Benzonatate Soft Capsules for Improving Adult Cough Symptoms
Brief Title: A Study on the Efficacy and Safety of Benzonatate Soft Capsules for Improving Adult Cough Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EY20170501
Record Dates: First submitted 2018-10-25; First posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-03

CONDITIONS: Cough
MeSH Terms: conditions — Cough | interventions — benzonatate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- benzonatate soft capsules group (Active Comparator)
  Interventions: Drug: Benzonatate 200 mg
- control group (Placebo Comparator)
  Interventions: Drug: blank control 0mg

INTERVENTIONS:
Drug: Benzonatate 200 mg — 200 mg/pellet, 1pellet/time, 3times/day
  Arms: benzonatate soft capsules group
Drug: blank control 0mg — 0 mg/pellet, 1pellet/time, 3times/day
  Arms: control group

SUMMARY:
The purpose of this study is evaluate the efficay and safety of benzonatate soft capsules for improving adult cough symtoms.

DETAILED DESCRIPTION:
The purpose of this study is evaluate the efficay and safety of benzonatate soft capsules for improving adult cough symtoms. The study was designed to be randomized, double-blind, placebo-controlled.Subjects were randomly assigned to the benzonatate soft capsule group and the placebo group on a 1:1 basis。According to the regulatory requirements, 200 cases were planned to be included. Considering that poor efficacy of the placebo control group might lead to shedding, a 10% increase in shedding was achieved, and 220 cases were finally determined, with 110 cases in each group.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18 and 75 years of age;
2. the onset time is more than 3 days and less than 8 weeks;
3. dry cough, the total score of cough symptom in day and night is greater than 4;
4. Willing to sign informed consent.

Exclusion Criteria:

1. allergic person or known to the test drug containing ingredients (including benzo, soybean oil, glycerin, gelatin) allergy;
2. the cough symptoms are caused by bronchial asthma, tuberculosis, pneumoconiosis, bronchiectasis, tumor and other diseases that have been clearly diagnosed.
3. coughers caused by drugs;
4. respiratory depression or airway obstruction;
5. patients with uncontrolled diabetes or hypertension;
6. having difficulty in swallowing or affecting drug absorption, such as active peptic ulcer and acute gastritis;
7. patients with severe hematopoietic system, nervous system, mental illness (including alcohol and substance abuse) or immunodeficiency diseases;
8. laboratory examination results are abnormal with clinical significance, among which: A.C r is higher than normal value; B.A LT and/or AST>2 times normal value upper limit (ULN).
9. women during pregnancy or lactation or women who are preparing for pregnancy or lactation during the trial;
10. in the first 3 months of screening, any other experimental drug treatment was accepted;
11. Failure to comply with test plans or other conditions that other researchers believe is not appropriate for the group.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
reducion of cough symptoms total scores | 7days
  The reduction of cough symptoms will be evaluated by comparative score index basal and final score

CONTACTS AND LOCATIONS:
Overall Officials: Cao Zhaolong, M.D., Principal Investigator — Peking University People's Hospital
Locations (14):
- China (14):
  - Beijing hospital, Beijing, Beijing Municipality
  - Beijing luhe hospital affiliated to capital medical university, Beijing, Beijing Municipality
  - Beijing pinggu district hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Second affiliated hospital of Harbin medical university, Harbin, Heilongjiang
  - Zhengzhou first people's hospital, Zhengzhou, Henan
  - Second Hospital of Xiangya, Changsha, Hunan
  - Affiliated hospital of Inner Mongolia medical university, Hohhot, Inner Mongolia
  - Inner Mongolia autonomous region people's hospital, Hohhot, Inner Mongolia
  - First hospital of jilin university, Changchun, Jilin
  - Jilin Province People's Hospital, Changchun, Jilin
  - Affiliated Zhongshan Hospital Dalian University, Dalian, Liaoning
  - First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Central hospital of yangpu district, Shanghai, Shanghai, Shanghai Municipality